CLINICAL TRIAL: NCT06648252
Title: Healing Minds: Biofeedback and Breathing Practices in Children and Adolescents With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoskinson Health and Wellness Clinic (Industry)
Responsible Party: Principal Investigator, Inara McMaster, Director of Pediatrics, Hoskinson Health and Wellness Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRANY IRB File #24-10-211-1498
Record Dates: First submitted 2024-10-16; First posted 2024-10-18 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Two-arm Randomized and Controlled Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healing Minds (Experimental): Ten weekly treatments of Heart Math Biofeedback and Breathing Practices
  Interventions: Behavioral: Healing Minds Biofeedback and Breathing Practices Intervention
- Control (No Intervention): Waiting List Delayed Intervention

INTERVENTIONS:
Behavioral: Healing Minds Biofeedback and Breathing Practices Intervention — The study participant will attend ten weekly Healing Minds sessions at the Hoskinson Health and Wellness Clinic. The parent (s) or guardian will accompany the study participant and follow along with the cues during the weekly session. Each session will be approximately 60 minutes. The principal investigator/pediatrician or trained and certified health care or research staff member will deliver the intervention. Biofeedback will be implemented based on the Heart Math Protocol. Breathing practices will include a variety of yoga and qi gong techniques.
  Arms: Healing Minds

SUMMARY:
The objective of this research proposal is to examine the combined effects of an integrative approach including biofeedback and breathing practices (Healing Minds) on severity of Attention Deficit Hyperactivity Disorder (ADHD) in youth 6-18 years of age. The investigators hypothesize that ADHD severity will be significantly reduced and Heart Rate Variability (HRV) increased after participation in the 10-week intervention. The investigators also propose that ADHD severity in those patients with prescribed medication but poorly-controlled ADHD will demonstrate the greatest improvement compared to those not prescribed medication and those who have well-controlled ADHD. Our specific aims are as follows:

AIM I. Conduct a randomized, placebo-controlled trial (RCT) to examine the effects of a 10-week integrative intervention (Healing Minds) that includes Heart Math Biofeedback and Breathing Practices on ADHD severity and HRV in children and adolescents 6-18 years of age diagnosed with ADHD (N=40). Participants randomized to placebo will be placed on a delayed intervention waiting list and will receive the 10-week Healing Minds intervention afterwards.

Hypothesis I: ADHD severity will be significantly reduced and HRV increased following the 10-week Healing Minds Intervention in children and adolescents, 6-18 years of age diagnosed with ADHD compared to a placebo condition

AIM Ia. Observe the effects of the Healing Minds intervention in the following sub-groups of youth:

ADHD without medication (well versus poorly controlled) ADHD with medication (well versus poorly controlled) Hypothesis Ia: Participants without medication will experience a significantly greater reduction in ADHD severity compared to those with medication. Poorly controlled participants with medication will experience the greatest reduction in ADHD severity.

AIM Ib. Explore the effects of the intervention on related mental health conditions:

PTSD Anxiety Resilience

DETAILED DESCRIPTION:
Attention-Deficit Hyperactivity Disorder (ADHD) affects 2.8% of adults and 5.9% of youth worldwide, and is more prevalent in males compared to females. There are both genetic and environmental risks for developing ADHD. As such, the condition is an epigenetic disorder with a complex pathophysiology that includes numerous biological pathways. Numerous co-morbidities are associated with ADHD including obesity, asthma, diabetes mellitus, and somatic disorders. Individuals diagnosed with ADHD are more likely to attempt and complete a suicide attempt. Chronic illnesses associated with ADHD are shown to develop early in life and track into adulthood. Thus, ADHD is a significant public health issue. The Healing Minds intervention will be implemented by a trained and certified pediatrician, health care or research staff member to children and adolescents diagnosed with Attention Deficit/Hyperactivity Disorder (ADHD). The proposed study will determine if the intervention is safe and effective compared to a placebo condition. The Healing Minds intervention includes a biofeedback component and breathing practices. Biofeedback is a type of mind-body technique used to control body functions such as heart, lung and muscle responses. Biofeedback uses therapeutic techniques that aim to help study participants gain more awareness and control over certain physiological functions in their bodies. It involves the use of electronic monitoring equipment to provide real-time information about physiological processes such as heart rate, heart rate variability and muscle tension. This information is then provided back to the study participant, allowing participants to learn how to consciously regulate these processes. During the sessions parents are expected to attend and participate. Study participants and parents will have access to a video that provides instructions for placement of the Heart Math single small ear lobe or finger sensor. Breathing Practices include alternate nostril, qi gong and other breathing practices. Biofeedback and breathing practices will be employed to help the study participants to: 1) Improve attention and focus by training the participants to regulate brainwave patterns and improve concentration, 2) Develop emotional regulation skills, helping study participants become more resilient in the face of stressors, 3) Control physiological responses can contribute to overall emotional well-being.

ELIGIBILITY:
Inclusion Criteria:

* 6-18 years
* Male and female children and adolescents
* Confirmed diagnosis of ADHD using the DSM-5-TR criteria

Exclusion Criteria:

* Severe, uncontrolled mental illness including depression, panic disorders
* Suicidal ideology
* Psychosis
* Severe, uncontrolled, autonomic nervous system or metabolic disorders including hypertension, diabetes, hypotension, autoimmune disease, or any condition that would limit their participation in the intervention
* Disorders involving severe impairments of memory or neurological conditions such as seizures
* Pregnant or nursing females may not participate because of some of the tests that are required for the study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2024-07-08 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
ADHD Severity | Baseline and Ten Weeks
  The Conner's Abbreviated Parents Rating Scale
ADHD Severity | Baseline and Ten Weeks
  The Conner's Abbreviated Teacher Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Inara McMaster, MD, Principal Investigator — Hoskinson Health and Wellness Clinic
Locations (1):
- Hoskinson Health and Wellness Clinic, Gillette, Wyoming, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McMaster, I., Hoskinson, W., Thompson, T., Stone, K., Sothern, M,, Pasam, H., Karanam, N., Missikpode, C., Dhar, S. Safety, Feasibility, Child and Parent Perceptions following Biofeedback and Breathing Practices in Children with Attention Deficit Hyperactivity Disorder: The Healing Minds Study, Journal of Clinical and Translational Science (abstract), in press.